CLINICAL TRIAL: NCT05149105
Title: Efficiency of Using Argon Plasma Coagulation in Weight Regain in Patients Following Gastric Bypass. Monocentric, Comparative, Randomized, Open Study.
Brief Title: Efficiency of Using Argon Plasma Coagulation in Weight Regain in Patients Following Gastric Bypass
Acronym: ARG-BP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint-Gregoire Private Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A02992-37
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Bariatric Surgery Candidate
MeSH Terms: interventions — Argon Plasma Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APC intervention (Experimental): In addition to multidisciplinary care (standard care), patients benefit from an Argon Plasma Coagulation (APC) intervention at D0.
  The APC intervention should be repeted at Month 2 and Month 4.
  Interventions: Procedure: Argon plasma coagulation
- Control (No Intervention): Patients are treated according to standard care (multidisciplinary care).

INTERVENTIONS:
Procedure: Argon plasma coagulation — On D0, in the operating room, argon plasma coagulation will be performed around the perimeter of the anastomosis for a period of 5 to 10 min under general anesthesia. The removal of the catheter and the endoscope will be carried out under control. Patients will be kept under surveillance the night following the procedure. A liquid diet will be prescribed for 10 days. The follow-up will be carried out on an outpatient basis with a control endoscopy at 2 months, followed by a new procedure in the event of an anastomosis larger than 1.5 cm. A new endoscopic check will be carried out at 4 months if an argon plasma coagulation was performed during the previous check, with a third and last argon plasma coagulation if an anastomosis of more than 1.5 cm persists. The number of procedures will therefore be a maximum of 3. A control endoscopy will be performed at one year for the final control of the anastomosis.
  Arms: APC intervention

SUMMARY:
Among the techniques of bariatric surgery, the gastric Y bypass according to Roux (RYGB) allows greater weight loss and more lasting over time than sleeve gastrectomy and gastric banding. However, around 20% of patients will regain weight within 24 months after surgery. Among the many mechanisms that lead to weight regain, we can mention distension of the gastric pouch and gastro-jejunal anastomosis. A reoperation is then necessary. Argan plasma coagulation intervention (APC) by endoscopy allows to reduce the caliber of the gastro-jejunal anastomosis. The aim of the study is to show the efficacy of APC associated with multidisciplinary medical management and to compare it with multidisciplinary medical management alone in weight regain of patients.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 65 years old.
* Have had a gastric bypass in Y more than 2 years ago
* Have a weight regain of more than 10% of the lowest weight after the first intervention.
* Have benefited from a multidisciplinary medico-psychological reassessment.
* Understand the interest of the study and agree to long-term follow-up.
* Agree to be included in the study and have signed a consent form in a free and informed manner.
* Be affiliated with health insurance.
* For female patients of childbearing potential, have an effective method of contraception

Exclusion Criteria:

* Presence of a disease unrelated to obesity that is life-threatening.
* Pregnancy or wish to become pregnant within the year.
* "Breastfeeding" patients
* Female patients of childbearing age and unable or unwilling to use an effective method of contraception
* Presence of an unhealed gastric ulcer or stenosis of the gastrointestinal anastomosis
* Presence of a psychiatric pathology compromising the proper understanding of the study or patient under guardianship or guardianship.
* Patient not understanding French or unable to give consent.
* Patient already included in a study or in conflict of interest with this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of the percentage change (loss) in excess weight from Day 0 to Month 12 between the 2 arms | Day 0 (before the intervention) and Months 12 (one year after Day 0)
  The percentage of excess weight loss (PEP%) will be measured according to the formula: PEP% = weight loss in kg * 100 / excess of initial weight. The initial excess weight is defined as the baseline weight - ideal weight.

CONTACTS AND LOCATIONS:
Locations (1):
- CHP Saint-Grégoire, Saint-Grégoire, France

IPD SHARING:
Plan to Share IPD: Undecided